CLINICAL TRIAL: NCT06232278
Title: Long-term Results of Percutaneous Left Atrial Closure at Brest University Hospital.
Brief Title: Long-term Results of Percutaneous Left Atrial Closure at Brest University Hospital (CLAPOT)
Acronym: CLAPOT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0255 - CLAPOT
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Cardioembolic Stroke; Left Atrial Appendage Thrombosis; Anticoagulant-induced Bleeding
Keywords: Left atrial appendage occlusion · WATCHMAN · AMPLATZER Amulet · Atrial fbrillation · Stroke · Echocardiography · Cardiac computed tomography angiography
MeSH Terms: conditions — Atrial Fibrillation; Embolic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial Fibrillation represents an important risk of cardioembolic stroke. In more than 90% of cases, thrombus originate in the left atrial appendage. Therefore guidelines recommend the anticoagulation of patients with atrial fibrillation and a significant cardioembolic risk, predicted by the CHA2DS2VASc score.

However, serious bleeding complications may definitively contraindicate the use of anticoagulants.

For those patients, percutaneous Left Atrial Appendage Occlusion (LAAO) has became a recommended alternative to prevent the thrombus formation and reduce the risk of cardioembolic events.

In the CHU of Brest, more than 120 patients have been treated with LAAO for the last 8 years with two different occluder devices : WATCHMAN®, Boston Scientifc and AMPLATZER Amulet®, Abbott Laboratories.

This retrospective longitudinal observational study named CLAPOT (CHU of Brest' Left Atrial Appendage Percutaneous Occlusion Treatment) aims to evaluate the long term results of this procedure for effectiveness and safety and to compare the results between the two devices (Watchman and Amplatzer).

ELIGIBILITY:
Inclusion Criteria:

* Major
* Non opposition
* All patients with non-valvular atrial fibrillation and a definitive contraindication to anticoagulants who underwent left atrial appendage occlusion in the CHU of Brest between December 2014 and August 2023

Exclusion Criteria:

* Minor
* Patients under tutorship or curatorship
* Formulated opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with non-valvular atrial fibrillation and a definitive contraindication to anticoagulants who underwent left atrial appendage occlusion in the CHU of Brest between December 2014 and August 2023
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of left atrial appendage occlusion with both devices WATCHMAN®, Boston Scientifc and AMPLATZER Amulet®, Abbott Laboratories | From 15 February 2024 to 15 April 2024
  Effectiveness is assessed by a composit endpoint that combines transient ischemic attack (TIA)/stroke, systemic embolism, cardiovascular mortality or All-cause mortality

SECONDARY OUTCOMES:
Safety of left atrial appendage occlusion (LAAO) with both devices WATCHMAN®, Boston Scientifc and AMPLATZER Amulet®, Abbott Laboratoriesleft atrial. | At 8 weeks
  The safety is defined as occurrence of events related to the device (device embolization, the presence of visible thrombus on the surface of the device, significant peri-device leak) and events related to the procedure (serious pericardial effusion requiring drainage, intracranial or gastrointestinal bleeding or other major bleeding requiring transfusion)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement